CLINICAL TRIAL: NCT02808832
Title: Development of an HPV Vaccine and Cervical Cancer Screening Provider Intervention
Brief Title: An HPV Vaccine Provider Intervention in Safety Net Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: Vanderbilt University (Other); Matthew Walker Comprehensive Health Center (Unknown); Memphis Health Center (Unknown); Southside/Dodson Avenue Community Health Centers (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U54CA153708 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Human Papillomavirus; Uterine Cervical Neoplasms
Keywords: Human papillomavirus (HPV) vaccine; Cervical cancer screening; Provider intervention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational materials (Experimental): 5-minute video and information sheet with a list of suggested questions to ask the provider
  Interventions: Behavioral: Educational materials
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Educational materials — 5-minute video and information sheet with a list of suggested questions to ask the provider
  Arms: Educational materials

SUMMARY:
The purpose of this study is to develop, deliver and evaluate a provider intervention for mothers and their children to encourage receipt of the human papillomavirus (HPV) vaccine in the children and appropriate cervical cancer screening in the mothers.

DETAILED DESCRIPTION:
In this study the investigators utilized Community Based Participatory Research approaches in combination with our previous and ongoing research, patient and provider education materials available from professional organizations, and qualitative information obtained from provider in-depth interviews and parent/daughter focus groups to develop a provider intervention to encourage receipt of the HPV vaccine, and appropriate cancer screening in African Americans and Hispanics. A focus of the study was the formation of a Community Advisory Board (CAB) which provided input into the development and modification of the provider intervention. Safety net clinics in Nashville and Memphis served as intervention sites, and in Chattanooga and Nashville (Meharry) served as control sites. Mothers and children at the intervention sites viewed a 5-minute video in the exam room during any visit type before seeing the provider, and received an information sheet with a list of suggested questions to ask the provider. Mothers and children at the control sites received usual care. The selected study sites identified cervical cancer screening as a priority area based on the needs assessments conducted as part of the Meharry Medical College Community Health Center-Community Network Program (CHC-CNP). The investigators conducted pre- and post-intervention quantitative surveys with mothers and their children to evaluate whether the provider intervention was effective in improving HPV vaccination coverage, and cervical cancer screening rates. The investigators abstracted medical records and have indicated this in the HIPAA privacy form. After conducting pre- and post-intervention surveys and abstracting medical records, the investigators found that increasing HPV vaccine uptake requires more intensive, multicomponent interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being seen as a pediatric patient at a study clinic on the day of enrollment
* Self-identified African American or Hispanic
* Aged 9-18 years (mother accompanying child to clinic visit had no age limit)
* Had received no doses of HPV vaccine or received one shot and was overdue for the second dose (three or more months after the first dose was given) prior to the clinic visit

Exclusion Criteria:

* Already having received two or more doses of HPV vaccine
* Mother or female guardian (referred to as "mother" henceforth) not accompanying the child
* Plans to move away from the clinic catchment area within the next 12 months
* Not completing the baseline assessment prior to entering the exam room
* Mother not providing or unable to give consent
* Child not giving assent.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2010-09; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of children participants who completed the 3-dose HPV vaccine series | 12 months
  Although completion of the 3-dose HPV vaccine series is recommended within 6 months, the investigators measured completion within 12 months.

SECONDARY OUTCOMES:
Number of mother participants who received appropriate cervical cancer screening | 12 months
  Cervical cancer screening is no longer recommended annually so the investigators measured receipt of a Pap smear as needed within a 12 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Sanderson, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanderson M, Canedo JR, Khabele D, Fadden MK, Harris C, Beard K, Burress M, Pinkerton H, Jackson C, Mayo-Gamble T, Hargreaves MK, Hull PC. Pragmatic trial of an intervention to increase human papillomavirus vaccination in safety-net clinics. BMC Public Health. 2017 Feb 2;17(1):158. doi: 10.1186/s12889-017-4094-1. PMID 28153042